CLINICAL TRIAL: NCT05786404
Title: A Randomized, Open-label, Pilot Study to Evaluate the Fecal Microbiota Transplantation (FMT) in the Treatment of Ulcerative Colitis
Brief Title: Study to Evaluate the Fecal Microbiota Transplantation (FMT) in the Treatment of Ulcerative Colitis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Andrew Dupont, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-23-0016
Record Dates: First submitted 2023-03-13; First posted 2023-03-27 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Active Ulcerative Colitis (UC)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: PRIM-DJ2727 - FROZEN (Experimental)
  Interventions: Drug: PRIM-DJ2727 - FROZEN
- Experimental: PRIM-DJ2727 - CAPSULES (Experimental)
  Interventions: Drug: PRIM-DJ2727 - CAPSULES

INTERVENTIONS:
Drug: PRIM-DJ2727 - FROZEN — Patients with active UC will receive induction dose of 100 grams of stool via frozen retention enema, Fecal Microbiota Transplantation (FMT) product manufactured as PRIM-DJ2727-FROZEN administered in clinic. This consists of microbiota suspension from well-screened donors. Twice filtered fecal microbiota product diluted in saline to 500 mL containing 100g of study drug will be administered as frozen enema induction dose
  Arms: Experimental: PRIM-DJ2727 - FROZEN
Drug: PRIM-DJ2727 - CAPSULES — Patients with active UC will receive induction dose of 100 grams of stool in orally administered enteric-coated capsules Fecal Microbiota Transplantation (FMT) product manufactured as PRIM-DJ2727-CAPSULES.These capsules consists of microbiota from well-screened donors. The induction dose of enteric-coated capsules will be derived from 100 grams stool.
  Arms: Experimental: PRIM-DJ2727 - CAPSULES

SUMMARY:
The study is to evaluate the safety, feasibility, and preliminary efficacy of frozen FMT delivery via retention enema compared to lyophilized powder given in oral capsules as induction FMT in subjects with active UC. This study will also determine changes in microbiome (diversity and genera) and proportion of antibody-coated microbiota from baseline to after completion of FMT.

DETAILED DESCRIPTION:
Studies have shown that microbiota disturbances occur in patients with ulcerative colitis (UC). This study will evaluate safety and preliminary efficacy of microbiota replacement treatment in active UC, and changes in microbiome (diversity and genera) and proportion of antibody-coated microbiota from baseline to after completion of FMT. Studies have shown that microbiota disturbances occur in patients with ulcerative colitis (UC). This study will evaluate safety and preliminary efficacy of microbiota replacement treatment in active UC, and changes in microbiome (diversity and genera) and proportion of antibody-coated microbiota from baseline to after completion of FMT.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of active UC defined on clinical grounds (Partial Mayo score ≥ 3 with each subscore >1)
* Sexually active male and female subjects of childbearing potential must agree to use an effective method of birth control during the study.
* Female subjects of childbearing potential must have a negative urine Qualitative Human Chorionic Gonadotropin(HCG)pregnancy test at enrolment and on the Week 1, Day 1 of the Treatment prior to administration of study drug.
* Willing and able to sign an informed consent form and attend all study-related clinic visits, assessments, and follow-up phone calls.
* Subject has an attending physician who will provide the non-FMT care.

Exclusion Criteria:

* Subjects with sever UC (Mayo score of >7)
* Unable to take retention enema or multiple capsules orally.
* Females who are pregnant, breastfeeding, or planning to become pregnant during the study.
* Receipt of systemic non-topical antibiotics within 14 days of treatment day 1.
* Positive results for active HIV, Hepatitis B, or Hepatitis C infections.
* History of recurrent Clostridium difficile infection or FMT in the past 6-months.
* History of other active gastrointestinal conditions such as irritable bowel syndrome, microscopic colitis, celiac disease, short gut syndrome, colostomy, colectomy, gastrointestinal fistulae or strictures, chronic parasitic infections, diverticulitis etc.
* Known history of bile acid diarrhea
* Compromised immune system (e.g. primary immune disorders or clinical immunosuppression due to a medical condition or medication e.g. taking oral prednisone >20 mg a day or prednisone-equivalent)
* History of active cancer and/or ongoing chemotherapy (superficial non-metastatic cancers and maintenance chemotherapy are permitted).
* History of use of an investigational drug within 90 days prior to the screening visit.
* History of significant uncontrolled systemic disease that in the opinion of the study investigator could interfere with study participation and/or objectives.
* Life expectancy of < 1 year.
* In the opinion of investigator, subject for any reason, should be excluded from the study.
* Absolute neutrophil count (ANC) < 500IU/mL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Disease severity as assessed by the Partial Mayo Score (PMS) for Ulcerative Colitis (UC) | week 5
  This is a 3 item questionnaire and each is measured from 0-3, for a maximum score of 9 a higher number indicating worse outcome
Change in fecal microbiota diversity and genera as assessed by sequencing | Baseline,end of treatment (4 weeks after baseline)
Change in proportion of antibody-coated microbiota as assessed by the antibiotic susceptibility test | Baseline,end of treatment (4 weeks after baseline)
Safety as assessed by the adverse events | 3 months after last dose
  Adverse events include death, life-threatening adverse event, hospitalization ≥ 24 hours, prolongation of existing hospitalization, substantial disruption of the ability to conduct normal life functions, congenital abnormally/birth defect, persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions or other important events that jeopardize the patient and may require medical or surgical intervention (e.g. allergic bronchospasm requiring intensive treatment)
Safety as assessed by the adverse events | 6 months after last dose
  Adverse events include death, life-threatening adverse event, hospitalization ≥ 24 hours, prolongation of existing hospitalization, substantial disruption of the ability to conduct normal life functions, congenital abnormally/birth defect, persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions or other important events that jeopardize the patient and may require medical or surgical intervention (e.g. allergic bronchospasm requiring intensive treatment)

SECONDARY OUTCOMES:
Change in quality of life as assessed by the Short Inflammatory Bowel Disease Questionnaire (SIBDQ) score | baseline, week 5, early termination(if applicable)
  This is a 10 item questionnaire and each is scored from 1(all of the time) to 7 (none of the time) for a maximum score of 70 a higher number indicating better quality of life
Change in anxiety and depression as assessed by the Hospital Anxiety and Depression Scale (HADS) | baseline, week 5, early termination(if applicable)
  This is a fourteen-item questionnaire to assess anxiety and depression. Seven items are related to anxiety symptoms and seven to depressive symptoms. Each item is coded from 0 to 3. The scores for anxiety and depression can therefore vary from 0 to 21, a higher number indicating worse outcome
Change in fecal microbiota diversity and genera as assessed by sequencing | Baseline,end of treatment (4 weeks after baseline), 6 months
Change in proportion of antibody-coated microbiota as assessed by the gut microbiota taxonomy by sequencing | Baseline,end of treatment (4 weeks after baseline), 6 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Herbert L DuPont, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No